CLINICAL TRIAL: NCT06168214
Title: Standard or Short-course Vonoprazan Non-bismuth Triple Therapy or High-dose Dual Therapy Versus Rabeprazole-bismuth Quadruple Therapy for Primary Helicobacter Pylori Eradication: A Single-center, Randomised, Controlled Trial.
Brief Title: Standard or Short-course Vonoprazan Non-bismuth Triple Therapy or High-dose Dual Therapy Versus Rabeprazole-bismuth Quadruple Therapy for Primary Helicobacter Pylori Eradication
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Han Ying, Prof, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJLL-KY-20230499
Record Dates: First submitted 2023-11-24; First posted 2023-12-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: the Eradication Rates of Helicobacter Pylori
Keywords: Helicobacter pylori ; Vonoprazan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Rabeprazloe+bismuth+amoxicillin+clarithromycin 14days (Active Comparator): 14D: PPI: Rabeprazole 10mg bid; B: bismuth potassium citrate240mg bid/ colloidal bismuth pectin 300mg bid/ colloidal bismuth tartrate 220mg bid; A:amoxicillin1000mg bid; C: clarithromycin 500mg bid.
  Interventions: Drug: Rabeprazloe+bismuth+amoxicillin+clarithromycin
- Vonoprazan+amoxicillin+clarithromycin 14 days (Experimental): 14D: V: vonoprazan 20mg bid; A:amoxicillin1000mg bid; C: clarithromycin 500mg bid.
  Interventions: Drug: Vonoprazan+amoxicillin+clarithromycin 14 days
- Vonoprazan+amoxicillin+clarithromycin 7 days (Experimental): 7D: V: vonoprazan 20mg bid; A:amoxicillin1000mg bid; C: clarithromycin 500mg bid.
  Interventions: Drug: Vonoprazan+amoxicillin+clarithromycin 7 days
- Vonoprazan+tetracycline+furazolidone 14 days (Experimental): 14D: V: vonoprazan 20mg bid; T: tetracycline 500mg tid; F: furazolidone 100mg bid.
  Interventions: Drug: Vonoprazan+tetracycline+furazolidone 14 days
- Vonoprazan+tetracycline+furazolidone 7 days (Experimental): 7D: V: vonoprazan 20mg bid; T: tetracycline 500mg tid; F: furazolidone 100mg bid.
  Interventions: Drug: Vonoprazan+tetracycline+furazolidone 7 days
- Vonoprazan+amoxicillin+furazolidone 7 days (Experimental): 7D: V: vonoprazan 20mg bid; A:amoxicillin1000mg tid; F: furazolidone 100mg bid.
  Interventions: Drug: Vonoprazan+amoxicillin+furazolidone 7 days
- Vonoprazan+amoxicillin+tetracycline 14 days (Experimental): 7D: V: vonoprazan 20mg bid; A:amoxicillin1000mg tid; T: tetracycline 500mg tid.
  Interventions: Drug: Vonoprazan+amoxicillin+tetracycline 14 days
- Vonoprazan+amoxicillin 7 days (Experimental): 7D:V: vonoprazan 20mg bid; A:amoxicillin1000mg tid.
  Interventions: Drug: Vonoprazan+amoxicillin 7 days
- Vonoprazan+amoxicillin 14 days (Experimental): 14D:V: vonoprazan 20mg bid; A:amoxicillin1000mg tid.
  Interventions: Drug: Vonoprazan+amoxicillin 14 days

INTERVENTIONS:
Drug: Rabeprazloe+bismuth+amoxicillin+clarithromycin — PBAC: 14D: PPI: Rabeprazole 10mg bid; B: bismuth potassium citrate240mg bid/ colloidal bismuth pectin 300mg bid/ colloidal bismuth tartrate 220mg bid; A:amoxicillin1000mg bid; C: clarithromycin 500mg bid.
  Arms: Rabeprazloe+bismuth+amoxicillin+clarithromycin 14days
Drug: Vonoprazan+amoxicillin+clarithromycin 14 days — VAC14: 14D: V: vonoprazan 20mg bid; A: amoxicillin1000mg bid; C: clarithromycin 500mg bid.
  Arms: Vonoprazan+amoxicillin+clarithromycin 14 days
Drug: Vonoprazan+amoxicillin+clarithromycin 7 days — VAC7: 7D: V: vonoprazan 20mg bid; A: amoxicillin1000mg bid; C: clarithromycin 500mg bid.
  Arms: Vonoprazan+amoxicillin+clarithromycin 7 days
Drug: Vonoprazan+tetracycline+furazolidone 14 days — VTF14: 14D: V: vonoprazan 20mg bid; T: tetracycline 500mg tid; F: furazolidone 100mg bid.
  Arms: Vonoprazan+tetracycline+furazolidone 14 days
Drug: Vonoprazan+tetracycline+furazolidone 7 days — VTF7: 7D: V: vonoprazan 20mg bid; T: tetracycline 500mg tid; F: furazolidone 100mg bid.
  Arms: Vonoprazan+tetracycline+furazolidone 7 days
Drug: Vonoprazan+amoxicillin+furazolidone 7 days — hVAF: 7D: V: vonoprazan 20mg bid; A: amoxicillin1000mg tid; F: furazolidone 100mg bid.
  Arms: Vonoprazan+amoxicillin+furazolidone 7 days
Drug: Vonoprazan+amoxicillin+tetracycline 14 days — hVAT: 14D: V: vonoprazan 20mg bid; A: amoxicillin1000mg tid; T: tetracycline 500mg tid.
  Arms: Vonoprazan+amoxicillin+tetracycline 14 days
Drug: Vonoprazan+amoxicillin 7 days — hVA7: 7D: V: vonoprazan 20mg bid; A: amoxicillin1000mg tid.
  Arms: Vonoprazan+amoxicillin 7 days
Drug: Vonoprazan+amoxicillin 14 days — hVA14: 14D: V: vonoprazan 20mg bid; A: amoxicillin1000mg tid.
  Arms: Vonoprazan+amoxicillin 14 days

SUMMARY:
The goal of this clinical trial is to compare eradication rates of Helicobacter pylori in patients aged 18-70 years with first infection. The main questions it aims to answer are:

* Main indicators: the eradication rate of Helicobacter pylori for eradication.
* Secondary indicators: symptomatic relief rate at 2 weeks after treatment and 4 weeks after the end of treatment; compliance and adverse reactions during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years, regardless of sex; chronic gastritis, peptic ulcer or dyspeptic symptoms, clear Hp infection (positive 13C-urea breath test); voluntary Hp eradication treatment; women of childbearing age are required to use a medically desirable form of contraception during the trial and for 1 month after the trial.

Exclusion Criteria:

* Have contraindications to the study drug or are allergic to the study drug; have taken a PPI within 2 weeks and an antibiotic or bismuth within 4 weeks; pregnant and lactating women; and Have undergone upper gastrointestinal surgery; refluse to sign the informed consent document.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1404 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-11-25 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori | Helicobacter pylori eradication rate assessed 4-8 weeks after completion of treatment
  Evaluated by 13C/14C-urea Breath test results and/or monoclonal faecal antigen test results were assessed as negative for successful eradication and positive for negative for successful eradication, positive for failed eradication 13C/14C-urea breath test results and/or monoclonal faecal antigen test results, negative for successful eradication and positive for (assessed by 13C/14C-urea breath test results and/or monoclonal faecal antigen test results, negative for successful eradication, positive for failure).

SECONDARY OUTCOMES:
Incidence of adverse effects | 14 days of treatment, and 28 days after treatment
  According to the requirements of the "Drug Clinical Trial Management Code", the observation is carried out, and the adverse reactions of the patients during the administration of the drug are recorded. The severity, or intensity, of an AE refers to the extent to which an AE affects the subject' s daily activities. The intensity of the AE will be rated as mild (discomfort without influencing daily activities), moderate (discomfort partially influencing daily activities), or severe (discomfort with severe interruption with daily activities).
Treatment compliance | 7 or 14 days of treatment
  Adherence was analysed according to medication possession ratio (MPR), where taking less than 80% of study drug during any evaluation period or failure to review was considered poor adherence;
Symptom relief rate | 14 days of treatment, and 28 days after treatment
  Patients were classified as no change, remission, cure, or exacerbation based on changes in clinical symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Ying han, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes